CLINICAL TRIAL: NCT06552650
Title: Randomized Controlled Study to Evaluate the Effect of Early Exercise on Functional Restoration of Exercise and Surgical Outcomes After Breast Reconstruction
Brief Title: Evaluating the Effectiveness of an Early Exercise Program After Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2023-1146
Record Dates: First submitted 2024-02-28; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-02

CONDITIONS: Braest Cancer; Breast Reconstruction
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental)
  Interventions: Behavioral: Exercise
- Usual Care Group (Experimental)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Exercise — Four supervised exercise interventions after surgery: One exercise education session per week from postoperative day 5 through 1 month Subsequent home-based exercise: Home-based exercise recommendations from 1 month to 3 months post-surgery
  Arms: Exercise Group
Other: Usual Care — The full spectrum of patient care practices in which clinicians have the opportunity (which is not necessarily seized) to individualize care
  Arms: Usual Care Group

SUMMARY:
Breast reconstruction is an important step and option after mastectomy and can help improve the quality of life of breast cancer patients. Therefore, the proportion of patients undergoing breast reconstruction in conjunction with mastectomy is steadily increasing. Despite recent advances in less invasive techniques, postoperative movement restrictions are unavoidable, and these postoperative pain or functional limitations can last for months to years. Patients most often experience a decrease in shoulder function, which negatively impacts their physical function and is an important factor in their ability to perform activities of daily living. Early postoperative exercise has been proven to have positive results in promoting the recovery of shoulder function in breast cancer patient. However, there is a lack of research on the effectiveness of early postoperative exercise in the context of breast reconstruction. Therefore, this study aims to evaluate the effect of early postoperative exercise on patients' shoulder and trunk function after breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women between the ages of 19 and 70
2. Pathologically diagnosed with breast cancer
3. Scheduled to undergo unilateral or bilateral mastectomy and breast reconstruction

Exclusion Criteria:

1. Adult women age 70 and order who have been diagnosed with breast cancer
2. Had surgery or radiation therapy to the same side of the armpit
3. Scheduled to undergo or have undergone delyed breast reconstruction
4. Have breast cancer that has spread to other cancers or is metastatic
5. Deemed by the healthcare provider to have unmeasurable postoperative complications (seroma, laceration, lymphedema observed within 1 month of surgery)
6. Have problems reading or understanding Korean or have problems communicating with the researcher
7. Have difficulty exercising as judged by the healthcare provider

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder Range of Motion | "1 Day before surgery", "5 Days after Surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  Shoulder Range of Motion: Objectively measures shoulder range of motion (in degree) and measurements include shoulder flexion, abduction, internal rotation, external rotation and extension.
Shoulder Strength | "1 Day before surgery", "5 Days after Surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  Shoulder Strength: Objectively measures shoulder strength (in newton) and measurements include shoulder flexion, abduction, internal rotation, external rotation and extension.
Trunk Range of Motion | "1 Day before surgery", "5 Days after Surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  Trunk Range of Motion: Objectively measures trunk extension range of motion (in degree).
Trunk Strength | "1 Day before surgery", "5 Days after Surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  Trunk Strength: Objectively measures trunk flexion strength (in newton).

SECONDARY OUTCOMES:
Weight | "1 Day before surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  Weight (in kilograms) will be measured with InBody
BMI | "1 Day before surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  BMI (in kg/m²) will be measured with InBody
Body fat | "1 Day before surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  Body fat (in percentage) will be measured with InBody
Muscle mass | "1 Day before surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  Muscle mass (in kilograms) will be measured with InBody
Shoulder Pain and Disability | "1 Day before surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  DASH (Disabilities of the Arm, Shoulder, and Hand) questionnaires) questionnaires will be administered to asses shoulder pain and disability. Minimum value of 0, maximum value of 100, with higher scores indicating greater dysfunction
Postoperative Satisfaction after Breast reconstruction | "1 Day before surgery", "10-14 Days after surgery", "1 Month after surgery", "3 Months after surgery", "6 Months after surgery"
  Postoperative Satisfaction after Breast reconstruction: BREAST-Q questionnaires will be administered to assess postoperative satisfaction (satisfaction with breast, psychosocial well-being, and sexual well-being). Minimum value of 0 and a maximum value of 100, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Plastic Surgery, Yonsei University School of Medicine, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No